CLINICAL TRIAL: NCT00769054
Title: Lokal Infiltrations Analgesi Med Ropivakain 1 % Versus Placebo VED Vaginale Descensusoperationer: ET Prospektivt Randomiseret, Dobbeltblindet, Placebo- Kontrolleret Studie
Brief Title: Local Infiltration Analgesia With Ropivacaine in Posterior Vaginal Wall Prolapse:a Randomized, Double-Blind Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Billy B Kristensen, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H-C-2008-035
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2008-10

CONDITIONS: Vaginal Prolapse
Keywords: Postoperative pain; PONV
MeSH Terms: conditions — Uterine Prolapse; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Local Infiltration with Ropivacaine
  Interventions: Drug: Ropivacaine
- 2 (Placebo Comparator): Local Infiltration with Placebo
  Interventions: Drug: Isotonic NaCl

INTERVENTIONS:
Drug: Ropivacaine — Local Infiltration Analgesia with 1 % Ropivacaine
  Arms: 1
Drug: Isotonic NaCl — Local Infiltration with NaCl
  Arms: 2

SUMMARY:
The purpose of this study is to compare systematic local infiltration with ropivacaine or placebo in patients undergoing repair of posterior vaginal wall prolapse.

The hypothesis is that LIA technique is opioid-sparing and a better postoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* eligible for elective repair of posterior vaginal wall prolapse
* able to speak and understand Danish
* able to give informed consent

Exclusion Criteria:

* alcohol or medical abuse
* allergies to local anesthetics
* age < 18 yrs.
* intolerance to opioids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain during rest, coughing and ambulation | ½, 1, 2, 4, 8, 12 and 24 h postoperatively

SECONDARY OUTCOMES:
Postoperative Nausea and Vomitus | ½, 1, 2, 4, 8, 12 and 24 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Billy B Kristensen, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark